CLINICAL TRIAL: NCT06777173
Title: Clinical Study of Antiviral Therapy Combined With Novel Immunotherapy for Chronic Hepatitis B in Adults
Brief Title: Clinical Study of Antiviral Therapy Combined With Novel Immunotherapy for CHB in Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of Department, Beijing Ditan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023YFC2308105
Record Dates: First submitted 2024-11-24; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Chronic Hepatitis b; Immunotherapy
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): NAs combined with PegIFNa-2b therapy
  Interventions: Drug: Peg interferon alfa-2b

INTERVENTIONS:
Drug: Peg interferon alfa-2b — NA combined with Peg interferon alfa-2b
  Other Names: NA combined with Peg interferon alfa-2b

SUMMARY:
Establish a study cohort of adult chronic hepatitis B antiviral treatment based on the principle of responseguidedtreatment (RGT) corresponding to the child cohort, analyze the clinical cure factors of IC and IT stage adults chronic hepatitis B, and optimize the antiviral treatment plan. To determine the safety and efficacy of PD-1 antibody combined with Peg-FNa-2b in the treatment of adult NAs patients with CHB advantage.

DETAILED DESCRIPTION:
This research group established an adult randomized controlled study cohort corresponding to the children cohort: 1 immunetolerance (IT) and 1 immuneclearance (IC) antiviral treatment cohort, respectively according to 1: 1 Randomly divided into two intervention groups: nucleoside (acid) analogues (NAs) and NAs combined with pegylated interferon α-2b (PegIFNα-2b). 1 NAs treatment-advantaged population antiviral combined with novel immunotherapy cohort: PD-1 antibody, PegIFNα-2b and combination group were randomly enrolled 1:1:1, and the response guidance treatment plan was adjusted according to the response of patients during treatment, the HBsAg clearance rate at 24 weeks and 48 weeks of different optimal treatment groups was evaluated, the clinical curative characteristics and differences between children and adults were compared, and the key factors affecting clinical cure were screened. To determine the safety and efficacy of PD-1 antibody combined with Peg-FNa-2b in the treatment of adult NAs patients with CHB advantage.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old；
* Meet the 2022 Chronic Hepatitis B Guidelines definition of chronic HBV infection: HBsAg and/or HBVDNA positive >6 months;；
* Immune clearance period: HBeAg positive, HBVDNA positive, ALT>40U/L;
* Newly treated patients;
* Willing to sign informed consent

Exclusion Criteria:

* Patients with HAV, HCV, HEV infection and autoimmune liver disease; Pregnant and lactating women and patients who plan to give birth in the near future;
* Patients with cirrhosis or liver cancer indicated by imaging or liver hardness testing;
* A history of serious heart disease, including unstable or uncontrolled heart disease within the last 6 months;
* Have a mental illness or history of mental illness;
* Have uncontrolled seizures;
* Alcoholics or drug users who have not abstained;
* Have uncontrolled diabetes, hypertension, thyroid disease, retinopathy, autoimmune disease, etc.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
HBsAg clearance at 48 weeks. | 48weeks
  HBsAg clearance in enrolled patients at week 48.（The detection of serum HBV markers is carried out using a HBsAg quantitative Elecsys （Roche Diagnostics GmbH, German）, with a HBsAg quantitative detection limit of 0.05IU/mL.）

SECONDARY OUTCOMES:
Serum HBsAg clearance or conversion rates at week 24, week 72, and week 24 after drug withdrawal | 24 weeks,72 weeks
  Serum HBsAg clearance or conversion rates.（The detection of serum HBV markers is carried out using a HBsAg quantitative Elecsys （Roche Diagnostics GmbH, German）, with a HBsAg quantitative detection limit of 0.05IU/mL.）
HBeAg conversion rate at week 24, 48, 72 and 24 weeks after drug withdrawal | 24 weeks,48 weeks,72 weeks
  HBeAg conversion rate.（The detection of serum HBV markers is carried out using a HBsAg quantitative Elecsys （Roche Diagnostics GmbH, German）, with a HBsAg quantitative detection limit of 0.05IU/mL.）
The degree of serum HBsAg and HBeAg reduction from baseline at week 24, 48, 72 and 24 weeks after drug withdrawal | 24 weeks,48 weeks,72 weeks
  The degree of serum HBsAg and HBeAg reduction from baseline.（The detection of serum HBV markers is carried out using a HBsAg quantitative Elecsys （Roche Diagnostics GmbH, German）, with a HBsAg quantitative detection limit of 0.05IU/mL.）
The proportion of serum HBVDNA lower than the lower limit of detection at week 24, 48, 72 and 24 weeks after drug withdrawal | 24 weeks,48 weeks,72 weeks
  The proportion of serum HBVDNA lower than the lower limit of detection.（HBV DNA detection: Real time fluorescent quantitative PCR system is used for detection, with a detection limit of 10 IU/ml.）
Evaluation of drug safety during treatment | 36 months
  Evaluation of drug safety during treatment.(The rate of adverse reactions experienced by patients during medication use.)

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, Doctor, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan hospital, Beijing, China